CLINICAL TRIAL: NCT05047705
Title: Investigating Distress Tolerance in Adults With Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00298541
Record Dates: First submitted 2021-09-13; First posted 2021-09-17 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Tourette Syndrome; Tic Disorders; Tics
Keywords: Tourette Syndrome; Distress Tolerance; Premonitory Urge; Tic Disorders; Distress tolerance skill training
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distress Tolerance Skills Training (Experimental): Distress tolerance skills training is a multicomponent intervention drawn from third-wave cognitive-behavioral therapy (CBT) protocols.
  Interventions: Behavioral: Distress Tolerance Skills Training

INTERVENTIONS:
Behavioral: Distress Tolerance Skills Training — Individuals with TS will receive distress tolerance skill training. Therapeutic skill training will consist of 4 weekly 1-hour sessions. Skill training will occur either in-person or remotely via videoconferencing software. Sessions will focus on building participants' distress tolerance skills with strategies drawn from third-wave CBT.

SUMMARY:
Although behavior therapy is recognized as a first-line intervention for Tourette's Disorder (TD), less than 40% of adults with TD respond to this evidence-based treatment. Limited tolerance for aversive premonitory urges and affective states that accompany tics may be one likely factor that impedes behavior therapy outcomes. This study examines the relationship between distress tolerance and tic inhibition among adults with TD, and investigates the mechanism and effect of therapeutic skills training to enhance distress tolerance abilities. Findings will determine the optimal approach to enhance distress tolerance among adults with TD and ultimately lead to better behavior therapy outcomes.

DETAILED DESCRIPTION:
Tourette's Disorder and other persistent tic disorders collectively affect about about 1% of the population, cause significant distress, and functional impairment. Although behavior therapy is recognized as a first-line intervention for Tourette's Disorder (TD), less than 40% of adults with TD respond to this evidence-based treatment. Limited tolerance for aversive premonitory urges and affective states that accompany tics may be one likely factor that impedes behavior therapy outcomes. This study examines the relationship between distress tolerance and tic inhibition among adults with TD, and investigates the mechanism and effect of therapeutic skills training to enhance distress tolerance abilities.

ELIGIBILITY:
Participants will be eligible for participation if the following inclusion criteria are met:

* at least 18 years of age
* have moderate tic severity or greater as evidenced by a YGTSS Total Tic Score greater than 14 (>9 for adults with motor or vocal tics only)
* exhibit a tic frequency of at least one visible tic per minute
* be fluent in English
* have a total premonitory urge for tics scale (PUTS) total score greater than 17 at Visit 2
* have a total DTS score greater than 30 at Visit 2

Exclusion criteria for participants include:

* history of cardiovascular disorder
* history of fainting or seizures
* history of frostbite
* open cut or sore on hand to be immersed
* fracture to the limb to be immersed
* history of Reynaud's phenomenon
* inability to complete rating scales
* inability to attend study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Distress Tolerance Scale (DTS) | Within 1 week after completion of Distress Tolerance Skills Training
  The Distress Tolerance Scale is a 15-item self-report measure that measures the perceived capacity to tolerate distress from a multidimensional framework, including tolerance, appraisal, absorption, and regulation. Items are rated on a 1-5 Likert scale, and then summed. Score ranges from 15-75. Higher total scores indicate greater difficulty with tolerating distress.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale-Revised (YGTSS) | Within 1 week after completion of Distress Tolerance Skills Training
  The YGTSS is a clinician-rated semi-structured interview that measures tic symptom severity over the previous week. It consists of 10-items that assess different dimensions of tic severity for motor and vocal tics, which are rated on a 0-5 scale. The YGTSS produces a Total Tic Score (range: 0-50), with higher ratings indicating greater tic severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. McGuire, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No